CLINICAL TRIAL: NCT00092846
Title: A Consumer Use Study of OTC Lovastatin (CUSTOM): A 6-Month Consumer Behavior Study of the Lovastatin OTC Self-Management System
Brief Title: A 6-Month Consumer Behavior Study of a Self-Management System (0803-084)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0803-084; 2004_061
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Hypercholesterolemia
Keywords: High Blood Cholesterol Levels
MeSH Terms: conditions — Hypercholesterolemia | interventions — Lovastatin

INTERVENTIONS:
Drug: MK0803, lovastatin
Behavioral: Self-Management System

SUMMARY:
The purpose of this study is to evaluate the ability of patients with intermediate risk of heart disease to appropriately use a Self-Management System.

DETAILED DESCRIPTION:
The duration of treatment is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and understand English without assistance.
* For Males: Minimum age 45 years and Maximum age N/A (No limit).
* For Females: Minimum age 55 years and Maximum age N/A (No limit).

Exclusion Criteria:

* Pregnant or nursing
* Drug allergy

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2002-12-04 (Actual); Primary Completion 2003-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who make appropriate decision for self-management.

SECONDARY OUTCOMES:
Percentage of patients who make appropriate decision to discontinue therapy or consult with a physician; the incidence of adverse experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Melin JM, Struble WE, Tipping RW, Reynolds JM, Vassil TC, Levy SJ, Petrohoy TM, Midgette P, Hemwall EL, Levine JG, Irvin JD. A Consumer Use Study of Over-The-Counter lovastatin (CUSTOM). Am J Cardiol. 2004 Nov 15;94(10):1243-8. doi: 10.1016/j.amjcard.2004.08.007. PMID 15541238
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html